CLINICAL TRIAL: NCT01028456
Title: A Randomised Placebo Controlled Clinical Trial of Light Therapy for Medically Intractable Epilepsy.
Brief Title: Clinical Trial of Light Therapy for Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University College, London (Other)
Collaborators: Action Medical Research (Other)
Responsible Party: Mr Philip Diamond Senior Research Administrator, UCL
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09 H0716 68
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Epilepsy
Keywords: Seizures; Light Therapy
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100 lux (Placebo Comparator): 100 lux / 30 minutes day
  Interventions: Other: 100 lux
- Light Therapy 10,000 lux (Experimental): 10,000 lux / 30 minutes a day for 3 months
  Interventions: Other: Light Therapy

INTERVENTIONS:
Other: Light Therapy — 10,000 lux / 30 minutes a day
  Other Names: Diamond 4 light box
  Arms: Light Therapy 10,000 lux
Other: 100 lux — Placebo light
  Arms: 100 lux

SUMMARY:
This study is designed to investigate whether light therapy may be an effective treatment for some people with epilepsy. Light treatment is already an established treatment for depression. The chemical systems in the brain that are disrupted when someone becomes depressed, overlap with some of those that can be affected during some epileptic seizures. The investigators have designed this study to see whether light therapy may also lead to a decrease in seizures in people who have epilepsy.

The study will be a placebo controlled trial. This means that half of the participants will receive a therapeutic dose of light therapy from a light box, whilst the other half will only receive a placebo light treatment.

DETAILED DESCRIPTION:
The aim of this study is to investigate a new, non invasive treatment for epilepsy that may be useful as an adjunctive therapy for people whose seizures are poorly controlled with anti epileptic drugs. Light therapy is a well established treatment for some forms of depression. From the cellular level to epidemiological studies, there are numerous strands of evidence in the scientific literature that indicate that light therapy could be also an effective treatment for some people with epilepsy.

The proposed study is a randomised placebo controlled trial of light therapy. One hundred people with medically refractory epilepsy will be recruited. Participants will be randomised to receive either therapeutic or placebo doses of light therapy from an identical device for 30 minutes a day during the treatment phase of the study. The statistical power of this study design is >90% to detect a 25% reduction in seizure frequency during the treatment phase. Although this therapeutic approach is more likely to be palliative than curative, it represents a non invasive and relatively inexpensive add-on treatment option for a sub group of patients who may have reached the end of the road in other medical and surgical treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Medically intractable epilepsy
* Min 4 complex partial seizures/ month

Exclusion Criteria:

* Ability to give informed consent
* Underlying progressive neurological condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-04 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Number of seizures/month | 3 months

SECONDARY OUTCOMES:
Mood | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital for Neurology & Neurosurgery, London, London, United Kingdom

REFERENCES:
- [Derived] Baxendale S, O'Sullivan J, Heaney D. Bright light therapy for symptoms of anxiety and depression in focal epilepsy: randomised controlled trial. Br J Psychiatry. 2013 May;202(5):352-6. doi: 10.1192/bjp.bp.112.122119. Epub 2013 Mar 21. PMID 23520221
- [Derived] Baxendale S, O'Sullivan J, Heaney D. Bright light therapy as an add on treatment for medically intractable epilepsy. Epilepsy Behav. 2012 Jul;24(3):359-64. doi: 10.1016/j.yebeh.2012.04.123. Epub 2012 May 30. PMID 22658437